CLINICAL TRIAL: NCT05146492
Title: Pericardial Effusion From Acute Myocardial Infarction: Contributing Factors and Prognosis at One Year (EPERICARDIM)
Acronym: EPERICARDIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-A02590-57
Record Dates: First submitted 2021-11-25; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Acute Myocardial Infarction; Pericardial Effusion
MeSH Terms: conditions — Pericardial Effusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with acute myocardial infarction without pericardial effusion (Active Comparator)
  Interventions: Procedure: MRI
- Patient with acute myocardial infarction and pericardial effusion (Experimental)
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — MRI with gadolinium contrast media injection

SUMMARY:
This study aims to clarify, in patients with more or less abundant pericardial effusion in the acute phase of a myocardial infarction, the correlation between the existence of this effusion during the acute phase with clinical parameters, biological, angiographic, therapeutic and with transmurality, extent, microvascular obstruction and intra myocardial hemorrhage found on MRI made beyond one week and before the 3rd month of the constitution of the necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 90 years old
* Patient admitted to the acute or semi-recent phase (within the next fifteen days) of a myocardial infarction (primary or recurrent myocardial infarction) documented by a significant enzymatic release of troponin (threshold value at 100) in the course of: chest pain or shock, or flare-up of heart failure (left or global) or successfully resuscitated cardiac arrest, or paroxysmal ventricular arrhythmia with or without sus shift of the ST segment on the input trace, with or without Q wave of necrosis formed. This IDM may or may not be complicated by a more or less abundant pericardial effusion of more than 10 mm in the left parasternal, which may in the extreme be the cause of tamponade;
* Subject affiliated or beneficiary of a social security scheme;
* Patient having signed the free and informed consent.

Exclusion Criteria:

* Patient with a pericardial detachment of less than 10 mm, or only systolic;
* Patient who had a break-in during the primary angioplasty guide or complicated coronary dissection extravasation with secondary pericardial effusion;
* Patient with advanced chronic renal failure
* Patient unable to perform an MRI (with a defibrillator or pacemaker).
* Known allergy to contrast agents, in particular gadolinium
* claustrophobic patient;
* Protected patient: adult under guardianship or other legal protection, deprived of liberty by judicial or administrative decision;
* Pregnant or breastfeeding woman;
* Patient hospitalized without consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-01-19 (Estimated); Study Completion 2024-07-19 (Estimated)

PRIMARY OUTCOMES:
One-year mortality rate of patients with pericardial effusion | 1 year
  One-year mortality rate of patients with pericardial effusion

CONTACTS AND LOCATIONS:
Locations (1):
- Private Hospital of Parly II-Le Chesnay, Le Chesnay, France